CLINICAL TRIAL: NCT03538808
Title: Varenicline Pharmacological and Expectancy Effects on Medication Adherence (Balanced Placebo Design With Varenicline: Pharmacological and Expectancy Effects on Medication Adherence)
Brief Title: Balanced Placebo Design With Varenicline: Pharmacological and Expectancy Effects on Medication Adherence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Samantha Schiavon, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-300001404
Record Dates: First submitted 2018-05-15; First posted 2018-05-29 (Actual); Results first posted 2020-12-14 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-11

CONDITIONS: Medication Adherence
MeSH Terms: conditions — Medication Adherence | interventions — Varenicline

STUDY DESIGN:
Intervention Model Description: Balanced placebo design
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Therapeutic Dose Truth (Active Comparator): told therapeutic dose medication + received therapeutic dose medication
  Interventions: Drug: Varenicline
- Therapeutic Dose Deception (Placebo Comparator): told therapeutic dose medication + received placebo
  Interventions: Other: Placebo
- Low Dose Vareniclince Deception (Active Comparator): told low dose medication + received therapeutic dose medication
  Interventions: Drug: Varenicline
- Low Dose Placebo Deception (Placebo Comparator): told low dose medication + received placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Varenicline — Participants will be provided varenicline medication
  Arms: Low Dose Vareniclince Deception; Therapeutic Dose Truth
Other: Placebo — Participants will be provided placebo medication
  Arms: Low Dose Placebo Deception; Therapeutic Dose Deception

SUMMARY:
The current study will use the double-blind balanced placebo design to examine differences between expectancies versus the pharmacological effects of varenicline medication administered for two weeks to cigarette smokers. The double-blind balanced placebo design includes medication administration (active medication v. placebo) and medication information (told truth v. deception) resulting in four groups of smokers: (1) told therapeutic dose (TD) medication + received TD medication; (2) told TD medication + received placebo; (3) told low dose (LD) medication+ received TD dose medication; (4) told LD medication + received placebo. Ecological momentary assessments (EMA) in the form of Daily Dairies delivered via smartphone will assess real-time side effects, withdrawal symptoms, cigarettes smoked, medication use, and reasons for medication non-adherence.

DETAILED DESCRIPTION:
The current proposal will utilize the double-blind balanced placebo design to differentiate expectancies versus pharmacologic mechanisms of varenicline administered to varenicline naïve smokers seeking treatment (N = 80) for two-weeks. Race block randomization (controlling for baseline expectancies) will be used to randomize participants. The double-blind balanced placebo design includes a cross-balanced medication administration (active medication v. placebo) and instructional set (told truth v. deception) resulting in four groups of smokers seeking treatment (n = 20 for each): (1) told therapeutic dose (TD) medication + received TD medication; (2) told TD medication + received placebo; (3) told low dose (LD) medication+ received TD dose medication; (4) told LD medication + received placebo. Participants will be told they received low dose (rather than placebo) due to concerns that participants will not take a medication that they believe to be a placebo. Ecological momentary assessments (EMA) in the form of Daily Dairies delivered via smartphone will assess real-time side effects, withdrawal symptoms, cigarettes smoked, medication use, and reasons for medication non-adherence. The current proposal will test the following specific aims:

Specific Aim 1: Examine the main effects of instructional set and pharmacology. Hypothesis 1: Main effects for TD instructional set and active medication administration will result in reduced medication adherence compared with LD instructional set and placebo medication.

Specific Aim 2: Examine the interaction between instructional set and pharmacology. Hypothesis 2: There will be a synergistic (i.e., non-additive) effect between instructional set and pharmacology. Specifically, those assigned to the TD instructional set and active medication group will result in a 50% discontinuation compared to a 20% discontinuation in the TD instructional set and placebo medication group.

Exploratory Aim: Evaluate moderators of pharmacology and expectancy effects on medication adherence. First, we will conduct exploratory examination of baseline medication expectancies moderating the relationship between pharmacology and medication adherence. Second, we will conduct an exploratory evaluation of potential moderators (e.g., gender and race) of pharmacology and baseline medication expectancy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Smoking at least 5 cigarettes per day (cpd) for the past year
* A carbon monoxide (CO) >10ppm
* English speaking
* Must own a cellphone with SMS text capacity with Internet access OR daily use of email
* Must be varenicline naïve
* Express a desire to quit smoking

Exclusion Criteria:

* Living in a restricted environment (e.g., prison or jail facility, etc.)
* Pregnant or nursing
* Currently enrolled in a smoking cessation treatment program, using NRT products, or prescribed bupropion or varenicline
* Known allergy to varenicline
* History of kidney disease, dialysis or known kidney impairment
* Cognitive impairment or unstable psychiatric condition that interferes with the informed consent process (individuals stable on psychiatric medications will be included)
* Daily or exclusive use of other tobacco products
* Current suicidal or homicidal ideation or a suicidal attempt within the past 12 months
* History of stroke, heart attack, or seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2019-10-29 (Actual); Study Completion 2019-10-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: None, all participants that were enrolled in the study were randomized into one of the four conditions.
Groups:
- Therapeutic Dose/Varenicline: Participants were told they were provided with a therapeutic dose of varenicline and they received varenicline medication
- Therapeutic Dose/Placebo: Participants were told they received a therapeutic dose varenicline, but they received a placebo.
- Low Dose/Varenicline: Participants were told they received a very low dose varenicline, but they received a therapeutic dose varenicline.
- Low Dose/Placebo: Participants were told they received a very low dose varenicline, but they received a placebo.
Period: Overall Study
Arm/Group | Therapeutic Dose/Varenicline | Therapeutic Dose/Placebo | Low Dose/Varenicline | Low Dose/Placebo
Started | 20 | 20 | 20 | 20
Completed | 18 | 20 | 16 | 18
Not Completed | 2 | 0 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Therapeutic Dose/Varenicline | Therapeutic Dose/Placebo | Low Dose/Varenicline | Low Dose/Placebo | Total
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.15 (2.59) | 48.00 (2.59) | 45.00 (2.59) | 45.30 (2.59) | 46.86 (11.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 5 | 13 | 31
  Male | 15 | 12 | 15 | 7 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 20 | 20 | 19 | 19 | 78
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 10 | 10 | 10 | 10 | 40
  White | 9 | 10 | 10 | 10 | 39
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Stanford Expectations of Treatment Scale: Negative Subscale [Mean (Standard Deviation); unit: units on a scale] — The is a 3-item subscale scored on a 7-point scale ranging from 1 (strongly disagree) to 7 (strongly agree). This subscale measure has a minimum score of 3 and a maximum score of 21 with higher scores indicating greater negative expectancies (i.e., beliefs that varenicline will cause negative effects).
  units on a scale | 3.42 (0.34) | 3.2 (0.34) | 3.4 (0.34) | 3.3 (0.34) | 3.33 (1.48)

OUTCOME MEASURES:

1. Primary Outcome: Medication Adherence
Description: Self-reported medication adherence measured through a single item assessing medication compliance. The item is answered as "yes" (scored as 1) or "no" (scored as 0). This measure combines all responses from Day 1 through Day 13 of this study to provide a total measure of medication adherence ranging from 0% (missed all doses) to 100% (took every dose as prescribed). Higher scores indicate better outcomes (i.e., better adherence to medication).
Time Frame: Days 1 - 13
Measure: Number; unit: Percentage
Arm/Group | Therapeutic Dose/Varenicline | Therapeutic Dose/Placebo | Low Dose/Varenicline | Low Dose/Placebo
Number analyzed (Participants) | 18 | 20 | 16 | 18
Percentage | 85.36 | 86.79 | 81.93 | 86.09

2. Secondary Outcome: Medication Expectancies
Description: Medication expectancies will be measured through the Beliefs and Attitudes about Varenicline (BAV) scale which is a 6-item questionnaire adapted to assess varenicline expectancies. This measure is rated on a scale from 1 (not at all) to 5 (extremely). The measure has a minimum score of 6 and a maximum score of 30. Higher scores indicating better outcomes (i.e., stronger positive beliefs about using varenicline).
Time Frame: Baseline and Day 14
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Therapeutic Dose/Varenicline | Therapeutic Dose/Placebo | Low Dose/Varenicline | Low Dose/Placebo
Number analyzed (Participants) | 18 | 20 | 16 | 18
units on a scale | 3.56 [3.06 to 3.94] | 3.65 [3.12 to 4.18] | 3.50 [2.91 to 4.09] | 3.44 [2.89 to 4.00]

3. Other Pre Specified Outcome: Side Effects
Description: A 30-item self-report measure of the presence (or not) of symptoms commonly associated with varenicline side effects and nicotine withdrawal. Items are rated as "No" (scored as 0) or "Yes" (scored as 1). A total score was calculated to reflect the total number of reported side effects. This measure has a minimum score of 0 and a maximum score of 30. Higher scores indicate worse outcomes (i.e., greater frequency of experienced side effects).
Time Frame: Day 14
Measure: Mean (Standard Error); unit: Symptoms
Arm/Group | Therapeutic Dose/Varenicline | Therapeutic Dose/Placebo | Low Dose/Varenicline | Low Dose/Placebo
Number analyzed (Participants) | 18 | 20 | 16 | 18
Symptoms | 1.50 (0.57) | 3.40 (0.54) | 2.00 (0.61) | 1.89 (0.57)

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Therapeutic Dose/Varenicline | Therapeutic Dose/Placebo | Low Dose/Varenicline | Low Dose/Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 1/20 | 1/20 | 1/20 | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Therapeutic Dose/Varenicline (N=20) | Therapeutic Dose/Placebo (N=20) | Low Dose/Varenicline (N=20) | Low Dose/Placebo (N=20)
Depressed Mood (Psychiatric disorders) | 0 | 0 | 1 (1) | 0 — Pt depressed mood (denied any suicidal or homicidal ideations). Instructed to immediately stop medication and seek emergency services. Pt indicated that his symptoms ceased once he stopped the medication and was not in need of further treatment.
Nocebo Effect/Depressed Mood (Psychiatric disorders) | 0 | 0 | 0 | 1 (1) — Pt reported depressed mood and immediately stopped medication. Symptoms improved once she stopped the medication. It should be noted that this pt was assigned to the placebo condition (i.e., no varenicline was provided).
Nocebo Effect/Sexual Dysfunction (Renal and urinary disorders) | 0 | 1 (1) | 0 | 0 — Pt reported experiencing sexual dysfunction when taking the medication. Once medication was stopped, the symptoms ceased. It should be noted that this pt was assigned to a placebo condition (i.e., no varenicline medication was provided).
Nasal Polyp Removal (Surgical and medical procedures) | 1 (1) | 0 | 0 | 0 — Participant reported undergoing a surgery to remove a nasal polyp. This is not considered to be related to the study medication (varenicline).

LIMITATIONS AND CAVEATS:
(1) Reliance on self-report data, particularly for medication adherence, may have produced biased results with participants reporting higher adherence as an artifact of social desirability. (2) Although the primary outcome was to observe instances of nonadherence within the early initiation of varenicline, limiting the medication regimen to two weeks may have hindered observations in this study. (3) No information was collected related to the degree of severity for each reported side effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-05): https://cdn.clinicaltrials.gov/large-docs/08/NCT03538808/Prot_SAP_001.pdf